CLINICAL TRIAL: NCT01161004
Title: Pilot Study of EEG Signs of Awakening Secondary to Injection of Sugammadex: Evaluation by Recording Bispectral Index and NeuroSENSE (Prospective, Double-blind Study)
Brief Title: Recovery Effect of Sugammadex Measured by Bispectral and Neurosense Indices
Acronym: Sugarecovery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010/01
Record Dates: First submitted 2010-07-09; First posted 2010-07-13 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugammadex - Nacl 9/00 (Experimental): Sugammadex - Nacl 9/00:
  Patients will first receive sugammadex: 4 mg/kg when post tetanic count shows at least 1 or 2 responses; 2 mg/kg when Train of four shows at least 2 responses.
  In case of complete reversal of myorelaxation, total intravenous anesthesia is stopped and patients are allowed to awake.
  In the adverse case, patients wil receive Nacl 9/00 5 minutes after the first bolus of sugammadex.
  The study is finished 5 minutes after this second injection and care is let to the choice of the anesthesiologist in charge.
  Interventions: Drug: Sugammadex - Nacl 9/00
- Nacl 9/00 - sugammadex (Experimental): Nacl 9/00 - Sugammadex :
  Patients wil first receive Nacl 9/00. In case of complete reversal of myorelaxation, total intravenous anesthesia is stopped and patients are allowed to awake.
  In the adverse case, patients wil receive sugammadex 5 minutes after the first bolus of Nacl 9/00.
  Sugammadex is given as: 4 mg/kg when post tetanic count shows at least 1 or 2 responses; 2 mg/kg when Train of four shows at least 2 responses.
  The study is finished 5 minutes after the injection of sugammadex and care is let to the choice of the anesthesiologist in charge.
  Interventions: Drug: Nacl 9/00 - sugammadex

INTERVENTIONS:
Drug: Sugammadex - Nacl 9/00 — * Sugammadex: 4 mg/kg when post tetanic count shows at least 1 or 2 responses; 2 mg/kg when Train of four shows at least 2 responses.
  * Nacl 9/00: same volume as Sugammadex
  Other Names: Sugammadex: Bridion
  Arms: Sugammadex - Nacl 9/00
Drug: Nacl 9/00 - sugammadex — * Nacl 9/00: same volume as Sugammadex
  * Sugammadex: 4 mg/kg when post tetanic count shows at least 1 or 2 responses; 2 mg/kg when Train of four shows at least 2 responses.
  Other Names: Sugammadex: Bridion
  Arms: Nacl 9/00 - sugammadex

SUMMARY:
It has been demonstrated that antagonism of neuromuscular blockade (neostigmine 0.04 mg kg-1) affects depth of anaesthesia with an increase in bispectral index (mean maximal change of 7.1) and middle-latency auditory evoked potentials (mean maximal change of 9.7).

Sugammadex has a quicker and more complete effect than neostigmine. This study aims to demonstrate if sugammadex administration increases bispectral and neurosense indices of the depth of anesthesia while patients still receive propofol-remifentanil iv anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to receive general anesthesia with muscle relaxation

Exclusion Criteria:

* contra-indication to the administration of propofol, remifentanil, rocuronium and to the use of the Bispectral Index or NeuroSense monitor
* known drug allergy or hypersensitivity to a drug used in the study
* history of central brain injury
* patient treated with a psychotropic agent
* patient with a pacemaker
* severe renal insufficiency
* treatment by toremifene, flucloxacillin or fusidic acid in the preoperative or immediate postoperative period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
modification of bispectral and neurosenses indices following sugammadex injection | day 1 after anesthesia

SECONDARY OUTCOMES:
efficacy of sugammadex to reverse myorelaxation | day 1 after anesthesia
clinical signs of recovery after sugammadex injection | day 1 after anesthesia
residual myorelaxation in the post-anesthesia care unit | day 1 after anesthesia
score of White and Song during the three first postoperative hours | day 1 after anesthesia
duration of stay in the postanesthesia care unit | day 1 after anesthesia
occurence of explicit memorisation | day 1 after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

REFERENCES:
- [Background] Vasella FC, Frascarolo P, Spahn DR, Magnusson L. Antagonism of neuromuscular blockade but not muscle relaxation affects depth of anaesthesia. Br J Anaesth. 2005 Jun;94(6):742-7. doi: 10.1093/bja/aei120. Epub 2005 Mar 18. PMID 15778268
- [Derived] Le Guen M, Roussel C, Chazot T, Dumont GA, Liu N, Fischler M. Reversal of neuromuscular blockade with sugammadex during continuous administration of anaesthetic agents: a double-blind randomised crossover study using the bispectral index. Anaesthesia. 2020 May;75(5):583-590. doi: 10.1111/anae.14897. Epub 2019 Dec 5. PMID 31808151